CLINICAL TRIAL: NCT00432367
Title: The Effectiveness, Cost and Cost Effectiveness of Intermittent Preventive Treatment or Screening and Treatment of Malaria in Pregnancy Among Women Using Long Lasting Insecticide Treated Bed Net: a Randomised Controlled Trial.
Brief Title: Intermittent Preventive Treatment (IPTp) Versus Rapid Diagnostic Testing (RDT) and Treatment of Malaria in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kwame Nkrumah University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMP_REG04; HKT-GMP
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2014-02

CONDITIONS: Malaria; Anaemia; Pregnancy
Keywords: Malaria in pregnancy; Case management; Screening; RDT; IPTp; Amodiaquine; Artesunate
MeSH Terms: conditions — Malaria; Anemia | interventions — Amodiaquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): OptiMAL® antigen screening and treatment with SP plus LLIN
  Interventions: Drug: Amodiaquine plus artesunate combination; sulphadoxine-pyrimethamine
- 2 (Experimental): OptiMAL® antigen screening and treatment with AQ+AS plus LLIN
  Interventions: Drug: Amodiaquine plus artesunate combination; sulphadoxine-pyrimethamine
- 3 (Active Comparator): SP-IPTp plus LLIN
  Interventions: Drug: Amodiaquine plus artesunate combination; sulphadoxine-pyrimethamine

INTERVENTIONS:
Drug: Amodiaquine plus artesunate combination; sulphadoxine-pyrimethamine — Eligible women will be allocated randomly to one of three groups and treated as follows:
  Arm 1 (OptiMAL® antigen screening and treatment with SP plus LLIN group) - a woman in this will receive 1500mg/75mg (S/P) administered at the ANC as single dose on enrollment if her screening test is positive.
  Arm 2 (OptiMAL® antigen screening and treatment with AQ+AS plus LLIN) - a woman in this will receive 300mg of AQ and 100mg co-administered two times a day for 3 days if her screening test is positive. The first dose is observed on enrolment day at the ANC.
  Arm 3 (SP-IPTp plus LLIN group) - a woman in this will receive 1500mg/75mg (S/P) administered at the ANC as single dose on enrollment as recommended by national policy.
  All enrolled women will be given one long lasting insecticide treated bed net each for use.

SUMMARY:
Among the best practices recommended for malaria control during pregnancy is ensuring effective case management of malaria illness. However, this is often not practiced because (1) malaria infection in pregnancy is often asymptomatic, (2) peripheral parasitaemia may be absent even when the placenta is heavily parasitized, (3) implementing diagnosis and treatment of malaria within a routine antenatal service may be difficult and (4) antimalarial treatment options available to pregnant women are limited due to resistance to chloroquine(CQ) and sulfadoxine-pyrimethamine(SP0 and paucity of safety and efficacy data on other antimalarial drugs in pregnancy, particularly artemisinin combination treatments (ACT). Therefore the commonest recommended practice in pregnancy is the administration of SP as intermittent preventive treatment (SP-IPTp). However, the effectiveness of SP-IPTp has been questioned because parasite resistance to SP is spreading rapidly across sub-Saharan Africa.

This is a three-arm open label randomised control non-inferiority trial of insecticide-treated nets(ITN) plus rapid diagnostic test(RDT) screening, and treatment with SP or amodiaquine plus artimisinin(AQ+AS) versus ITN plus IPTp using SP. It is to be carried out in pregnant women of all parities presenting at enrolling antenatal clinics with a gestation of 16 to 20 weeks at their first booking. The key objectives are to demonstrate that (1) the prevalence of severe anaemia (Hb < 8g/dl) at 34 to 36 weeks of gestation (2) the prevalence of low birth weight (BW < 2500g) at delivery or within 72 hours after delivery (3) the prevalence of placenta parasitaemia and (4) the incidence of serious and non-serious adverse events in the ITN plus RDT screening and treatment arm are not greater than those in the ITN plus IPTp arm. Alongside the clinical assessments, health care cost assessments will be done to determine the cost-effectiveness of the two delivery strategies measured as cases of severe maternal anaemia averted.

DETAILED DESCRIPTION:
General objective To show that the long-lasting insecticide-treated nets(LLIN)///// plus RDT screening and treatment strategy is not inferior to LLIN plus SP-IPTp in reducing the burden of malaria during pregnancy.

Specific objectives Primary

1. To demonstrate that the prevalence of severe anaemia (Hb < 8g/dl) at 34 to 36 weeks of gestation in the LLIN plus RDT screening and case management arm is not greater than that in the LLIN plus IPTp arm.

Secondary

1. To demonstrate that the prevalence of low birth weight (BW < 2500g) at delivery or within 72 hours after delivery in the LLIN plus RDT screening and case management arm is not greater than that in the LLIN plus IPTp arm.
2. To demonstrate that the prevalence of anaemia (Hb < 11g/dl) at 34 to 36 weeks of gestation in the LLIN plus RDT screening and case management arm is not greater than that in the LLIN plus IPTp arm.
3. To demonstrate that the prevalence of placental parasitaemia in the LLIN plus RDT screening and case management arm is not greater than that in the LLIN plus IPTp arm.
4. To demonstrate that the incidence of spontaneous abortions, intrauterine deaths/stillbirths, neonatal and maternal mortality and developmental delays in the LLIN plus RDT screening and case management arm is not greater than that in the LLIN plus IPTp arm.
5. To demonstrate that the cost per case of (1) severe maternal anaemia averted (2) maternal anaemia averted (3) peripheral malaria averted and (4) placenta malaria averted is not higher in the LLIN plus RDT screening and case management arm than in LLIN plus SP-IPTp arm.

Sample size The prevalences of severe anaemia at delivery and low birth weight have been shown to be 12% and 5.7% respectively among Gambian multigravidae who received varying doses of SP-IPT (Mbaye et al. 2006). In the absence of local data from the proposed study site, we estimate that the prevalences of severe anaemia in the third trimester and low birth weight will be 12% and 6% respectively in the LLIN +SP-IPTp arm of this study, similar to that in the Gambian population.

For trial planning we have set a non-inferiority margin of 5%. This means we would consider the LLIN + RDT screening with SP or AQ+AS treatment options to be inferior to the LLIN +SP-IPTp option if the prevalence of severe anaemia at 34 to 36 weeks is 5% greater in the LLIN+RDT with SP or AS+AQ treatment arm than that is observed in the LLIN+SP-IPT arm. Since we expect the prevalence of severe anaemia in the LLIN +SP-IPTp arm would be 12%, we need 887 women per arm to detect a 5% difference between the two study arms at 95% significance with 90% power. Considering a 20% dropout rate we need 1110 women per arm.

Setting a non-inferiority margin of 5% seems clinically and statistically relevant; and yields a sample size that makes the execution of the study feasible within the time frame and with the resources available. Choosing a smaller margin than 5% may be too tight requiring large sample size of over 2000 per arm which might not be feasible and achievable within the time frame; a larger margin than 5% may be too liberal to compare the public health impact of these interventions.

We estimate that 925 women per arm can show with 90% power at 95% significance level and accounting for a 20% dropout rate, that the prevalence of low birth weight associated with the LLIN + RDT screening with or without SP or AQ+AS treatment is no worse than LLIN + SP-IPTp by a margin of 4%.

Since, a sample size of 1110 per arm is adequate to detect any effects of the interventions on both birth weight and maternal Hb, a total of 3330 pregnant women will be recruited into this study.

Study Design A three-arm open label randomised control non-inferiority trial of RDT screening with or without treatment with SP or AQ+AS versus IPTp using SP as follows: -

1. OptiMAL® antigen screening and treatment with SP plus LLIN
2. OptiMAL® antigen screening and treatment with AQ+AS plus LLIN
3. SP-IPTp plus LLIN

Study site and population The study will be conducted in the Ejisu-Juaben and Sekyere East districts of the Ashanti Region of Ghana. Enrolment will be done simultaneously at the antenatal clinics of the Effiduase and Juaben district hospitals and a sub district health centre in each of the districts. The Effiduase and Juaben hospitals have 50 and 40 beds respectively and provide all basic medical services including adult medicine, paediatrics, surgery and obstetrics and gynaecology. They run weekly antenatal clinic sessions and together they register an average of 220 new pregnant women per month. The sub district health centres (at Kwaso and Kumawu) are manned by qualified medical assistants and midwives. Together they register an average of 80 new pregnant women per month. All health facilities in the study districts including the proposed enrolling clinics offer SP-IPT to pregnant women following the MoH guidelines. Pregnant women in their second or third trimester diagnosed with malaria are treated with AQ+AS as recommended by the MoH at these facilities. The study population will comprise pregnant women presenting at the hospital's antenatal clinic with a gestation of 16 to 24 weeks at their first booking.

Enrolment Procedures

A schematic profile of the study is shown in Figure 1. All study women will be recruited from weekly antenatal clinic sessions held at the study sites over a period of one and half years. Three teams of midwives and their assistants put together and trained by the principal investigator (PI) will assist the PI and research teams to conduct the recruitment during antenatal clinic hours. The standard operating procedures at the clinic will be as follows:

1. Randomise pregnant women reporting at the ANC who consent to participate in the study into three arms: an IPTp arm, RDT screening and SP case management arm and RDT screening and AQ+AS case management arm. Distribute LLIN to eligible pregnant women in all arms.
2. Obtain blood for baseline investigations including haemoglobin level, thin and thick blood films for malaria parasite counts and, filter paper blood spots.
3. Assess all pregnant women in the RDT and treatment groups clinically and obstetrically prior to OptiMAL® dipstick screening; for those parasitaemic offer SP or AQ+AS and ingestion of first dose observed directly at the ANC. Encourage the women to regularly sleep under the bed nets provided and take their daily doses of iron and folic acid tablets.
4. For women in the RDT and treatment groups who are negative offer only daily doses of iron and folic acid tablets and encourage them to regularly sleep under the bed nets provided.
5. Women in the IPTp group will receive SP and ingestion will be directly observed at the ANC according to the national guideline. Encourage the women to regularly sleep under the bed nets provided and take their daily doses of iron and folic acid tablets.
6. Women who decline participation in the study will receive SP-IPTp according to the national guideline.

Antenatal Follow-Up Procedures

1. Day 7: Women receiving SP or AQ+AS treatment will be followed up actively on the day 7 post treatment to assess any adverse events during the week post treatment.
2. At 6 months: repeat SP-IPT for women in the IPT arm and treat women in the case management arm with SP or AQ+AS if they are RDT positive. Women in the case management arm with negative RDT would receive only haematinics. Ask all study women to regularly sleep under bed nets provided.
3. At 8 months: repeat SP-IPT for women in the IPT arm and treat women in the case management arm with SP or AQ+AS if they are RDT positive. Women in the case management arm with negative RDT would receive only haematinics. Ask all study women to regularly sleep under bed nets provided.
4. At 34 to 36 weeks: actively follow up women to sample blood by finger prick for haemoglobin measurements, slide smears for malaria parasite counts and filter paper blood spots.
5. Unscheduled visits: Women presenting with a history of fever during an unscheduled visit will be tested for malaria parasites. If they are found to be parasitaemic, they will be deemed to be a treatment failure and will be given quinine as rescue medication.
6. All pregnant women will receive haematinics packs at each of the follow ups.

Delivery and Postpartum Follow-up

1. The midwives will record all birth weights and note any stillbirths and perinatal deaths.
2. Midwives will record all congenital deformities for verification and confirmation by a clinician.
3. Visits will be made toall women and babies at 6 to 8 weeks post-delivery to obtain reports of any neonatal deaths or other adverse events.
4. At 6 weeks post-partum, if a woman has peripheral parasitaemia she will be treated with SP and followed up for parasite clearance on days 14 and 28 post-treatment. If there is no parasite clearance on day 14 and/or day 28 a course of rescue medication (quinine) will be given. This part of the study is necessary to assess the efficacy of SP to clear parasitaemia.

ELIGIBILITY:
Inclusion Criteria:

* Her pregnancy is confirmed at 16 to 24 weeks at their first booking.
* She is willing to participate and complete the test schedule, and has given informed consent.
* She is willing to have supervised delivered at maternity units in the district.
* She lives within the study district.

Exclusion Criteria:

* She has a past obstetric and medical history that will adversely affect the interpretation of outcomes such as repeated stillbirths and eclampsia.
* She has a haemoglobin level below 5.0 g/dl.
* She has malaria that is severe enough to require parenteral medication.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3333 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of severe maternal anaemia (Hb < 8g/dl) at 34 to 36 weeks of gestation. | At 34 to 36 weeks of gestation

SECONDARY OUTCOMES:
Prevalence of low birth weight (BW < 2500g) at delivery or within 72 hours of delivery. | At delivery or within 72 hours of delivery.
Prevalence of maternal anaemia (Hb < 11g/dl) at 34 to 36 weeks of gestation. | At 34 to 36 weeks of gestation
Prevalence of placenta parasitaemia. | At delivery
Incidence of post-intervention malaria cases | Anytime after enrolment and prior to delivery
Proportions of congenital anomalies in live births among the intervention groups stratified by gestation, gravidity, parity and age. | At delivery
Proportions of spontaneous abortions, intrauterine death, stillbirths, neonatal and maternal mortality and pre-term deliveries. | Anytime after enrolment and prior to delivery
Cost per severe maternal anaemia averted. | Anytime after enrolment and prior to delivery
Cost per (non-severe) maternal anaemia averted. | Anytime after enrolment and prior to delivery
Cost per peripheral malaria case averted. | Anytime after enrolment and prior to delivery
Cost per placental malaria averted. | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Harry Tagbor, DrPH, Principal Investigator — School of Medical Sciences, KNUST, Kumasi, Ghana; Brian Greenwood, MD, Principal Investigator — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Jane Bruce, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Edmund Browne, PhD, Principal Investigator — School of Medical Sciences, KNUST, Kumasi, Ghana
Locations (1):
- Juaben Government Hospital, Juaben, Ashanti Region, Ghana

REFERENCES:
- [Derived] Tagbor H, Bruce J, Agbo M, Greenwood B, Chandramohan D. Intermittent screening and treatment versus intermittent preventive treatment of malaria in pregnancy: a randomised controlled non-inferiority trial. PLoS One. 2010 Dec 28;5(12):e14425. doi: 10.1371/journal.pone.0014425. PMID 21203389